CLINICAL TRIAL: NCT00581399
Title: A Prospective, Randomized, Multicenter Clinical Study on the High Vacuum Body Cavity Drainage Systems Following Open Heart Surgery
Brief Title: A Randomized Multicenter Clinical Study On the High Vacuum Body Cavity Drainage System Following Open Heart Surgery
Acronym: NO-NUMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: hs#2006-5196
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2011-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Artery Disease; Heart Valve Disease
Keywords: Open heart surgery; Cardiopulmonary Bypass; Coronary Artery Bypass Grafting; Chest Tube; Valve Replacement; Valve Repair
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NO-NUMO Chest Tube (Experimental): The NO-NUMO™ High Vacuum Body Cavity Drainage System consist of disposable NO-NUMO™ body cavity drainage tubes, disposable Vario™ fluid management canisters Vario™ portable vacuum pump
  Interventions: Device: NO-NUMO™ High Vacuum Body Cavity Drainage System
- Standard Chest Tube (Active Comparator): Classic PVC Chest Tube
  Interventions: Device: PVC Chest Tube

INTERVENTIONS:
Device: NO-NUMO™ High Vacuum Body Cavity Drainage System — (1) disposable NO-NUMO™ body cavity drainage tubes, (2) disposable Vario™ fluid management canisters and (3) Vario™ portable vacuum pump
  Arms: NO-NUMO Chest Tube
Device: PVC Chest Tube — Standard PVC Chest Tube Sizes 14-36 French
  Arms: Standard Chest Tube

SUMMARY:
The purpose of this study is to compare a new high vacuum pressure chest drainage system (NO-NUMO™) with the standard low vacuum pressure drainage system already in use in cardiac surgeries. The new system uses smaller diameter drainage tubing to remove blood from the chest after open heart surgery. This is less painful to the patient and should help the patient to breathe better after operation. Preliminary data suggests that the high vacuum suction is effective and practical, and could actually reduce the amount of chest tube bleeding after surgery without compromising heart function. This new high vacuum drainage system was approved by the FDA in 2002. Subsequent testing at University of California, Irvine indicated that this unique system may allow the surgeon to predict excessive postoperative bleeding before the patient is transferred out of the operating room, thus adding safety, convenience, and cost effectiveness to their use.

DETAILED DESCRIPTION:
High vacuum chest drainage was once considered inadvisable because of a possible suction injury to soft tissues, such as the lungs or mediastinum. Wakabayashi showed that excessive suction force generated by a high vacuum pressure was related to the surface area of the suction applied to the tissues and not the vacuum pressure itself1&2. He postulated that suction injury to the lung would not occur if the suction force of a chest tube is below the capillary blood pressure of 30 - 35 torr2. Based on this theory, Wakabayashi developed a double-lumen chest drainage tube3 (Trade name NO-NUMO™) and its clinical use was approved by FDA4 in 2002. A prototype 7-5Fr double-lumen chest tube was successfully tested in laboratory animals and three patients1&2 and the safety of high vacuum chest drainage was proven in a large number of patients undergoing uncomplicated thoracoscopic surgeries2. The unique design of the new drainage tube is the small diameter double lumen tube with hundreds of tiny holes that allows rapid drainage without damaging effects of high suction over a limited surface area. High vacuum suction is available on wall units already in place in the OR and ICU beds. To adopt this system for clinical use, a high vacuum gauge was needed (most don't go beyond 200 torr) to monitor suction, and a high pressure battery powered vacuum pump for transport was necessary, so that drainage was maintained and blood clotting in the tube avoided during the period of prolonged transport from the OR and the setup in the ICU. Several brands of portable vacuum pumps on the market were evaluated before concluding that the Vario™ pump (Medela® Inc.) was superior. The maximal vacuum pressure that Vario pump can generate is 630 torr or 84 kPa which is equivalent to -857 cmH2O.

The NO-NUMO™ High Vacuum Body Cavity Drainage System consist of; (1) disposable NO-NUMO™ body cavity drainage tubes, (2) disposable Vario™ fluid management canisters and (3) Vario™ portable vacuum pump. We evaluated this new system, using a 13Fr triple-tube set for the mediastinal drainage, a 13Fr single-tube for the left pleural drainage and two 13Fr NO-NUMO tubes for the drainage of the lower extremity subcutaneous wounds following the harvesting of the saphenous veins. The tubing was connected to a disposable liner of a Medi-Vac™ (Cardinal Health, Inc.) suction canisters, which was connected to a Vario pump at 300 torr (= 40 kPa) in patients following open heart surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 18 year-old or older
2. Patients undergoing open heart surgery by means of a standard cardiopulmonary bypass
3. The surgical procedures accepted include:

   1. Coronary-artery-bypass grafting
   2. Valve replacement or repair, or a combination of both
   3. Excision of a left ventricular aneurysm
   4. Bentall procedure is included but we do not include those undergoing replacement of the aortic arch aneurysm, utilizing deep hypothermic circulatory arrest.
   5. We include both first time operation and re-do operations.
   6. Patients with insulin dependent diabetes mellitus are included. Those with chronic renal failure who are on a hemodialysis treatment will be included.
   7. Emergency CABG for unstable angina following acute myocardial infarction
4. Patients must agreed to participate and sign an Informed Consent Form before the surgical procedure

Exclusion Criteria:

1. Transmyocardial laser revascularization
2. Open heart surgery for congenital heart diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2006-09; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Milliken, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects admitted to UCI Medical Center and scheduled for cardiac surgery (Coronary Artery Bypass Graft [CABG] with or without Heart valve repair, Heart valve repair alone without CABG) were randomized to one of two study arms: High Vacuum Chest Tubes or Standard of Care Chest Tubes. The enrollment period was from July 2006 through May 2010.
Pre-assignment Details: Only subjects that met specific study inclusion/exclusion criteria were enrolled into the study.
Groups:
- No-NumoChest Tubes: High Vacuum Chest Tubes 13Fr for Pleural Drainage and 22Fr connected to a Vario High Vacuum Pump (Medela) for Mediastinal Space Drainage.
- Standard of Care Chest Tubes: Standard of Care 36 Fr Chest Tubes connected to a Pleur-evac Chest Drainage System for Mediastinal Space Drainage.
Period: Overall Study
Arm/Group | No-NumoChest Tubes | Standard of Care Chest Tubes
Started | 46 | 48
Completed | 46 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No-NumoChest Tubes | Standard of Care Chest Tubes | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 15 | 17 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 36 | 34 | 70
Region of Enrollment [Number; unit: participants]
  United States | 46 | 48 | 94

OUTCOME MEASURES:

1. Primary Outcome: Amount of Postoperative Bleeding
Description: The outcome is to measure the amount of postoperative bleeding in cardiac surgery patients from the time the chest is completely closed until the chest tube is pulled out.
Time Frame: 24-48 hours post surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | No-NumoChest Tubes | Standard of Care Chest Tubes
Number analyzed (Participants) | 46 | 48
mL | 868.9 (430.17) | 1467.6 (1224.3)

2. Secondary Outcome: Duration of Mediastinal Drainage
Description: The outcome to measure is the duration of the chest tubes inserted in the patient in hours. The time starts at the time the chest is completely closed and the end time when the chest tubes are pulled out of the patient's chest.
Time Frame: Immediate postoperative when the chest is completely closed to the time chest tubes are pulled out of the patient
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | No-NumoChest Tubes | Standard of Care Chest Tubes
Number analyzed (Participants) | 46 | 48
Hours | 44.57 (22.5) | 54.74 (32.5)

ADVERSE EVENTS:
Arm/Group | No-NumoChest Tubes | Standard of Care Chest Tubes
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 0/46 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes